CLINICAL TRIAL: NCT06270706
Title: A Phase 1a/1b Multicenter, Open-label Dose Escalation/Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Evidence of Antitumor Activity of PLN-101095 as Monotherapy and in Combination With Pembrolizumab in Adult Participants With Advanced or Metastatic Solid Tumors Who Have Disease Progression While on Pembrolizumab
Brief Title: A Phase 1 Study of PLN-101095 in Adults With Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pliant Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PLN-101095-ONC-101
Record Dates: First submitted 2024-01-26; First posted 2024-02-21 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-02

CONDITIONS: Metastatic Solid Tumor
Keywords: Advanced Solid Tumors Cancer; Head and Neck Squamous Cell Cancer; Colorectal Cancer; Urothelial Carcinoma; Gastro-esophageal Junction Cancers; Esophageal Cancer; Cervical Cancer; Hepatocellular Carcinoma; Renal Cell Carcinoma; Endometrial Cancer; Cutaneous Squamous Cell Carcinoma; Triple Negative Breast Cancer; Melanoma; Non-Squamous Cell Lung Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Colorectal Neoplasms; Carcinoma, Transitional Cell; Esophageal Neoplasms; Uterine Cervical Neoplasms; Carcinoma, Hepatocellular; Carcinoma, Renal Cell; Endometrial Neoplasms; Triple Negative Breast Neoplasms; Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 Dose Escalation: PLN-101095 given as monotherapy and in combination with Pembrolizumab (Experimental)
  Interventions: Drug: PLN-101095; Drug: Pembrolizumab
- Part 2 Dose Expansion: PLN-101095 in combination with Pembrolizumab (Experimental)
  Interventions: Drug: PLN-101095; Drug: Pembrolizumab

INTERVENTIONS:
Drug: PLN-101095 — PLN-101095
Drug: Pembrolizumab — Pembrolizumab

SUMMARY:
This is a Phase 1a/1b, dose-escalation/expansion, consecutive-cohort, open-label study to evaluate the safety, tolerability, PK, PD, and preliminary evidence of antitumor activity of PLN-101095 in combination with pembrolizumab (the study treatment regimen) in adult participants with advanced or metastatic solid tumors for which pembrolizumab is indicated but have documented disease progression (refractory [primary resistance]) or relapsed [secondary resistance]) after at least 3 months from the start of treatment with pembrolizumab.

The study will consist of 2 main parts:

* Part 1: Consecutive dose-escalation cohorts using a Bayesian optimal interval (BOIN) dose escalation design
* Part 2: Dose-expansion cohorts using Simon's 2-stage design

ELIGIBILITY:
Inclusion Criteria:

1. Has histologically or cytologically confirmed advanced solid tumor
2. Has an advanced or metastatic solid tumor (for which pembrolizumab is indicated) and have evidence of disease progression after treatment with pembrolizumab.
3. At least 1 measurable lesion, as defined by RECIST v1.1
4. Estimated survival of ≥3 months
5. No effective therapeutic options available (eg, has received standard of care or is intolerant of, refuses, or is not eligible for standard of care antineoplastic therapy)

Exclusion Criteria:

1. Any immune-related medical conditions that would put participants at greater risk when receiving pembrolizumab
2. Previous treatment with pembrolizumab <21 days prior to the first dose of combination therapy of pembrolizumab and PLN-101095
3. Received an immunotherapy other than pembrolizumab in the last 4 weeks prior to the first dose of PLN-101095
4. Received radiotherapy (RT) within 1 week for palliative bone-directed therapy and 4 weeks for all other types, prior to the first dose of PLN-101095
5. Received chemotherapy or other targeted therapies within 2 weeks prior to the first dose of PLN-101095
6. Received a cell therapy within the last 12 months prior to the first dose of PLN-101095
7. Known active central nervous system (CNS) metastases (brain and/or leptomeningeal metastases)
8. Pregnant or lactating female participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with treatment-emergent adverse events and serious adverse events per CTCAE Version 5.0. | Signing ICF until 16 weeks after end of study treatment regimen
Number of participants with a Dose Limiting Toxicity (DLT) defined as toxicities that meet predefined severity criteria, assess as having a suspected relationship to study drug, unrelated to disease, inter-current illness, or concomitant medications. | First dose to 35 days

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) to characterize the plasma pharmacokinetics (PK). | First dose until 10 weeks
Time to maximum observed concentration (Tmax) to characterize the plasma pharmacokinetics (PK). | First dose until 10 weeks
Area under the concentration-time curve over a dosing interval (AUC0-τ) to characterize the plasma pharmacokinetics (PK). | First dose until 10 weeks
Disease control rate (DCR) is defined by the proportion of participants who maintain disease control (iCR, iPR or iSD) per iRECIST Version 1.1. | Day 1 until end of study treatment regimen
Objective response rate (ORR) is defined by the proportion of participants with an iCR or iPR per iRECIST Version 1.1. | Day 1 until end of study treatment regimen

CONTACTS AND LOCATIONS:
Overall Officials: Pliant Therapeutics Medical Monitor, Study Director — Pliant Therapeutics, Inc.
Locations (5):
- United States (5):
  - Yale University, New Haven, Connecticut
  - South Texas Accelerated Research Therapeutics (START), Grand Rapids, Michigan
  - NEXT Austin, Austin, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Virginia, Fairfax, Virginia